CLINICAL TRIAL: NCT04431973
Title: Étude Post-marché, Prospective, Multicentrique, Ouverte, d'évaluation de la prothèse Totale d'épaule inversée Medacta Shoulder System.
Brief Title: Open-label, Prospective, Multicenter, Post-market Study to Evaluate the Reverse Medacta Shoulder System of Total Shoulder Prosthesis.
Acronym: MSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DR190289-MSS; 2019-A03228-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-05-13; First posted 2020-06-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shoulder prothesis (Experimental): Evaluate the performance of the Medacta Shoulder System total reverse shoulder prothesis
  Interventions: Device: Medacta Shoulder System

INTERVENTIONS:
Device: Medacta Shoulder System — Surgical placement of the Medacta Shoulder System prothesis on patients with pathologies requiring the insertion of a total reverse shoulder prothesis for primary omarthrosis, cuff tear arthropathy, massive cuff rupture or post instability arthropathy

SUMMARY:
The goal of this study is to evaluate the performance of the Medacta Shoulder System total reverse shoulder prosthesis, at 2 years of follow up, in patients who required this prosthesis for primary omarthrosis, cuff tear arthropathy, massive cuff tear or post instability arthropathy.

The main goal is to evaluate at 2 years post-operatively the shoulder function of patients. The secondary goals are to assess the rate of complications, the survival rate of Reverse Medacta Shoulder System, the positioning of the prosthesis,pthe behaviour of the bone in contact with the humeral stem, Patient satisfaction and evolution of shoulder function in patients at 3 months and 1 year post-surgery.

DETAILED DESCRIPTION:
This study is a prospective, national, multicenter, non-controlled, non-randomized study in order to evaluate outcomes of the MSS reverse prosthesis used for the management of primary osteoarthritis, cuff tear arthropathy, massive cuff tear, or post-instability arthroplasty.

Included patients, will have an oral and written information about the study, including the information note, during a preoperative visit. The surgeon will answer any questions that may arise and will collect their decision after sufficient time for the patient to reflect.

Patients participating in the research will be able to withdraw their consent and ask to stop the study at any time and for any reason. The investigator should document the reasons as fully as possible.

Patients will be followed according to the schedule below:

* V1 : Inclusion during a preoperative visit
* V2: Surgery maximum 4 months after inclusion
* V3: Follow-up visit at 3 months ± 1 month post-surgery
* V4: Follow-up visit at 12 months ± 2 months post-surgery
* V5: Follow-up visit between 24 months and 28 months post-surgery, marking the end of follow-up for the patient.

The surgical technique for implantation of the Reverse Medacta Shoulder System total shoulder prosthesis will be performed according to the MyShoulder pre-operative planning (without custom-made guides). All procedures will be performed with conventional instrumentation according to each surgeon's current practice. It is possible to use the BIO-RSA technique to reposition the pre-morbid glenoid center. The stem that will be used is the short stem (cementless) with PE angulation at 145°.

The following data will be collected at each of the 3 month, 1 year and 2 year :

* Post-operative complications as dislocation, glenoid loosening, infection, neurological damage, fracture.
* Survival of implants according to these definitions Revision: A procedure that removes all or part of the original configuration of the implant, one or more of the components except for the polyethylene insert* if it has been removed and restored Re-operation: Any surgical procedure that does not remove, modify or add any components to the system.
* Clinical examination: evaluation of post-operative mobility, Constant score. This examination corresponds to current practice.
* Medical Imaging: the results of the radiological examinations will be reviewed centrally by independent assessors. These evaluators will collect the available data from the radiographs of the AP view, axillary profile, or Neer/Lamy. The data from the scans will be analyzed by each investigator and by the software.
* Patient questionnaire If a follow-up visit is not made, the reason will be collected and noted in the patient record and on the CRF. The investigator will proceed to obtain the most exhaustive follow-up data possible
* The clinical examination will be replaced by the Self-Constant Questionnaire which will be sent to the patient for completion.
* The results of available radiological examinations will be collected.
* The patient questionnaires planned for the study (ISS score and OSS score) will be sent to the patient for completion.

A web-based data collection medium will be used for this study. All the information required by the protocol will be collected in a e-crf. It requires only an Internet connection and a browser. A help document for the use of this tool will be provided to the investigators.

Data management for the study will be handled by a CIC INSERM 1415 data-manager. The electronic case report form (eCRF) will be developed using Ennov Clinical® software. Data management will be done according to the standard operating procedures (edited in CIC INSERM 1415. The Clinical Research Assistant in charge of the study will be trained in the use of the eCRF, then will be in charge of the training of investigators. Data relating to post-operative radiological data will be entered on the eCRF directly by the independent assessors commissioned for the centralized review of radiological examinations.

Analyses will be performed with SAS Version 9.4 (or later). The statistical analysis will be performed according to a pre-established statistical analysis plan. Missing values will not be replaced by estimated values but will be considered as missing in the statistical analysis.

A statistical analysis report will be written integrating all the elements to be reported.

A clinical research assistant will ensure the rigourous conduct of the study, the collection of the data generated in writing, their documentation, recording and reporting, in accordance with the Promotion and Quality Control Unit of the Tours CHRU as well as the legal and regulatory provisions.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 87 ;
* Patient with one of the following diseases: primary omarthrosis, cuff tear arthropathy, massive cuff tear or post instability arthropathy;
* Patient in need of a total shoulder prosthesis;
* Patient affiliated with or beneficiary of a social security scheme;
* Patient who has given written informed consent for the study.

Exclusion Criteria:

* Patient with malignant diseases;
* Patient with known or suspected infections;
* Patient with neurological deficits that may affect shoulder function;
* Patient with known incompatibility or allergy to product materials;
* Patient with previous open shoulder surgery (fracture sequelae, plate or nail, revision ...), treated for fractures, or suffering from rheumatoid arthritis (this does not concern patients treated by arthroscopy, or bone block);
* Protected major patient;
* Vulnerable person according to article L1121-6 of the Public Health Code;
* Pregnant or breastfeeding woman or woman of childbearing age;
* Impossibility to follow the consultation schedule planned in the study (planned move or mutation, etc...).

Exclusion criteria :

* Patient with malignant diseases on the day of surgery;
* Patient with known incompatibility or allergy to product materials on the day of surgery;
* Patient with known or suspected infections on the day of surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder function by evaluation of Constant's Score | 2 years post surgery
  The main evaluation criteria is the rate of improvement of the Constant Score and preoperative and postoperative mobility (active external and internal rotation, elbow to body) at 2 years post surgery.

SECONDARY OUTCOMES:
Complication rate | At 2 years post surgery
  Assess the complication rate associated with the MSS prosthesis (safety of the prosthesis, safety of the prosthesis, etc.).
Survival implants | At 2 years post surgery
  Evaluate the survival of Reverse Medacta Shoulder System implants
Position of the prosthesis | At 3 months, 1 year and 2 years post-surgery.
  Evaluate the positioning of the prosthesis by radiological analysis
Bone behaviour | At 3 months, 1 year and 2 years post-surgery.
  Evaluation of bone behaviour in contact with the humeral stem
Subjective Shoulder Value | At 3 months, 1 year and 2 years post-surgery
  Assess patient satisfaction after surgery at 3 months, 1 year and 2 years post-surgery
Oxford Shoulder Score | At 3 months, 1 year and 2 years post-surgery
  Assess patient satisfaction after surgery at 3 months, 1 year and 2 years post-surgery
Shoulder function by evaluation of Constant's Score | At 3 months and 1 year post-surgery
  Evaluate the evolution of shoulder function in patients who received a Medacta Shoulder System reverse ETP with MyShoulder preoperative planning (without custom guides).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Chu Angers, Angers
  - Chu Rennes, Rennes
  - Clinique Mutualiste la Sagesse, Rennes
  - Polyclinique santé atlantique, Saint-Herblain
  - Chu Tours, Tours